CLINICAL TRIAL: NCT06328010
Title: An Observational Clinical Registry to Collect Safety and Efficacy Data on Wound Care Treatments From a Variety of Treatment Settings
Brief Title: Clinical Registry Collecting Real World Evidence on Wound Care Treatments
Acronym: SIDDX
Status: Enrolling by invitation | Type: Observational
Sponsor: Siddhey LLC (Industry)
Collaborators: Acesso Biologics (Unknown); New Horizon Medical Solutions (Network)
Responsible Party: Sponsor
Other Study IDs: SIDDXAC02
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-10

CONDITIONS: Wounds and Injuries; Burns; Mohs Surgery; Diabetic Foot Ulcer Mixed; Venous Leg Ulcer; Non-healing Wound; Trauma Injury; Injury and Wounds; Degloving Injuries; Pressure Ulcers, Bedsores, Decubitus Ulcer
Keywords: Wound; DFU - Diabetic Foot Ulcer; VLU - Venous Leg Ulcer; Post Surgical; Trauma; Chronic Wound; MOHS - Mohs Micrographic Surgery; Non-Healing Wound
MeSH Terms: conditions — Wounds and Injuries; Burns; Varicose Ulcer; Accidental Injuries; Degloving Injuries; Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wound Treatment: Interventions are at the discretion of treating clinicians and include standard and advanced wound therapies.
  Interventions: Combination Product: Various types of wound care treatments

INTERVENTIONS:
Combination Product: Various types of wound care treatments — Treatments including, but not limited to:
  * Hydrocolloid
  * Foam
  * Alginate
  * Hydrogel
  * Collagen
  * Antimicrobial (e.g., silver, iodine)
  * Film
  * Composite
  * Negative Pressure (NPWT)
  * Amniotic-based

SUMMARY:
The proposed registry Sponsor (Siddhey LLC) will collect data on various wound treatments in real life settings. Data collection will facilitate the analysis of the safety and efficacy of wound treatments.

DETAILED DESCRIPTION:
This clinical registry is an observational study to collect prospective and retrospective data on subjects' health, wounds and wound care procedures from medical centers, including skilled nursing facilities, hospitals, outpatient clinics, Home Health and any other medical environment where wounds are treated.

The registry will enroll data of up to 5000 subjects in up to 100 wound care locations. The dataset includes all wound and ulcer types. Investigators will follow Institutional standards for routine wound care practices. The study products supplied through this study will be applied to the wounds as an adjunct to the standard of care treatment.

ELIGIBILITY:
Inclusion Criteria

1. Subject is male or female ≥18 years of age.
2. Subject has an ulcer (Diabetic foot ulcer, Venous stasis ulcer, etc.), injury (trauma, post -surgical, MOHS treatment), Burns injury, and/or other acute/chronic wounds.
3. Subject has clinical documentation of no visible wound improvement in the wound after 4 weeks of standard of care therapy.
4. Study wound is a minimum of 1 cm2 at Visit 1.
5. The subject is able and willing to follow the protocol requirements.
6. The subject has signed the informed consent form.
7. Subject has adequate circulation to the affected extremity. Note: This will be confirmed by vascular perfusion assessment performed prior to enrollment, if clinically indicated per Institutional standard of care.

Exclusion Criteria

1. Subject has a known life expectancy < 1 year.
2. Subject has major uncontrolled medical disorders such as serious cardiovascular, renal, liver, or pulmonary disease, lupus, palliative care or sickle cell anemia.
3. Subject currently being treated for an active malignant disease or subjects with a history of malignancy within the wound.
4. Known contraindications to advance therapy tissues or products.
5. Subjects with a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids >10 mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the wound surface within one month prior to Visit 1.
6. Affected extremity requiring hyperbaric oxygen during the study or within 2 weeks of Visit 1.
7. Known HbA1c >12%.
8. Subjects who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with wounds/injuries
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage wound area reduction over time while receiving study product using wound imaging device software or measurement scale | Up to 12 weeks
  Analysis will be based on product type (e.g., hydrocolloid, amniotic-based, etc.) and wound type (e.g., DFU, VLU, etc.)
Incidence and severity of treatment-emergent adverse events (TEAEs), including serious adverse events (SAEs), adverse events (AEs) related to wounds, and device-related adverse events (DRAEs) | Up to 12 weeks
  Note: Analysis will be based on product type (e.g., hydrocolloid, amniotic-based, etc.) and wound type (e.g., DFU, VLU, etc.)

SECONDARY OUTCOMES:
Proportion of wounds achieving complete closure over time | Up to 12 weeks
Time to achieve complete wound closure while receiving study product | Up to 12 weeks
Assessment of patient reported wound-related pain using a numeric pain rating scale of 0 (no pain) to 10 (worst possible pain) during study product application | Up to 12 weeks

OTHER OUTCOMES:
Care setting analysis for each type of care setting, the number of wounds per type of wound and severity of wound per year | Up to 12 weeks
  example: 20 severe DFUs per year
Care setting analysis for the duration of stay of wound (weeks) per type of admission | Up to 12 weeks
Economic comparison of treatment cost of wounds treated with Advanced biological/synthetic grafts. versus wounds treated with other treatments using classifications of wound type and medical center | Up to 12 weeks
Incidence of infection | Up to 12 weeks
Incidence of wound recurrence | Up to 1 year
Number of treatment applications | Up to 12 weeks
Percentage of wounds that closed during study product application that had previous therapy failure | Up to 12 weeks
Proportion of subjects adherent to standard of care therapy | Up to 12 weeks
  example: compression or offloading compliance as determined by the Investigator at each study visit

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Pulse Cardiovascular Institute, Scottsdale, Arizona
  - Metro Foot & Ankle, Tempe, Arizona
  - Pima Foot and Ankle Surgery LLC, Tucson, Arizona
  - Signature Health Medical Group, Riverside, California
  - The Schottenstein Center, Hallandale, Florida
  - PerfectFeetCare Podiatry Centers, Hialeah, Florida
  - The Schottenstein Center, Miami, Florida
  - PerfectFeetCare Podiatry Centers, Miami, Florida
  - Wigley Feet, North Miami Beach, Florida
  - Rubin Foot & Ankle, Naperville, Illinois
  - The Rache Clinic, Las Vegas, Nevada
  - Richard C. Galperin, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Data collected and analyzed will be marketed to researchers and manufacturers.

REFERENCES:
- See also: Wound care management market overview, 2017, By GlobalData Healthcare — https://www.medicaldevice-network.com/comment/wound-care-management-market-overview-2017/
- See also: Advanced Wound Care Market by Product Type (Infection Management, Exudate Management, Active Wound Care, Therapy Devices), Application (Chronic Wounds and Acute Wounds), End User (Hospitals and Community Centers)... — https://www.alliedmarketresearch.com/advanced-wound-care-market